CLINICAL TRIAL: NCT06305754
Title: A Randomized, Open-label, Phase 3 Study of MK-2870 vs. Platinum Doublets in Participants With EGFR-mutated, Advanced Nonsquamous Non-small Cell Lung Cancer (NSCLC) Who Have Progressed on Prior EGFR Tyrosine Kinase Inhibitors
Brief Title: Sacituzumab Tirumotecan (MK-2870) Versus Pemetrexed and Carboplatin Combination Therapy in Participants With Epidermal Growth Factor (EGFR)-Mutated, Advanced Nonsquamous Non-small Cell Lung Cancer (NSCLC) Who Have Progressed on Prior EGFR Tyrosine Kinase Inhibitors (MK-2870-009)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2870-009; 2023-504910-31-00 (Registry Identifier: EU CT); U1111-1288-3804 (Registry Identifier: UTN); MK-2870-009 (Other: MSD); jRCT2071240041 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Histamine Antagonists; Histamine H2 Antagonists; Acetaminophen; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Unblinded Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab tirumotecan (Experimental): Participants receive 4 mg/kg sacituzumab tirumotecan via intravenous (IV) infusion every 2 weeks (Days 1, 15, and 29 of every 6-week cycle) until discontinuation criteria is met.
  Interventions: Biological: Sacituzumab tirumotecan; Drug: H1 Receptor Antagonist; Drug: H2 Receptor Antagonist; Drug: Acetaminophen (or equivalent); Drug: Dexamethasone (or equivalent); Drug: Steroid Mouthwash (dexamethasone or equivalent)
- Pemetrexed Plus Carboplatin (Active Comparator): Participants receive, via IV infusion, 500 mg/m2 pemetrexed every 3 weeks (Days 1 and 22 of every 6-week cycle) plus area under the curve (AUC) 5 mg/mL*min carboplatin every 3 weeks (Days 1 and 22 of every 6-week cycle for 4 doses), then 500 mg/m2 pemetrexed every 3 weeks until discontinuation criteria is met.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — 4 mg/kg via IV infusion
  Other Names: SKB264; MK-2870
  Arms: Sacituzumab tirumotecan
Drug: Pemetrexed — 500 mg/m^2 via IV infusion
  Arms: Pemetrexed Plus Carboplatin
Drug: Carboplatin — AUC 5 mg/mL*min via IV infusion
  Arms: Pemetrexed Plus Carboplatin
Drug: H1 Receptor Antagonist — Administered as rescue medication per approved product label
  Arms: Sacituzumab tirumotecan
Drug: H2 Receptor Antagonist — Administered as rescue medication per approved product label
  Arms: Sacituzumab tirumotecan
Drug: Acetaminophen (or equivalent) — Administered as rescue medication per approved product label
  Arms: Sacituzumab tirumotecan
Drug: Dexamethasone (or equivalent) — Administered as rescue medication per approved product label
  Arms: Sacituzumab tirumotecan
Drug: Steroid Mouthwash (dexamethasone or equivalent) — Administered as rescue medication per approved product label
  Arms: Sacituzumab tirumotecan

SUMMARY:
The purpose of this study is to evaluate sacituzumab tirumotecan versus pemetrexed in combination with carboplatin for the treatment of epidermal growth factor receptor (EGFR)-mutated advanced non-squamous non-small cell lung cancer (NSCLC). Participants in this study have NSCLC that has continued to progress on prior treatment with EGFR tyrosine kinase inhibitors (TKIs).

The primary hypotheses of this study are that sacituzumab tirumotecan is better than platinum-based doublet chemotherapy (pemetrexed and carboplatin) in regard to progression-free survival (PFS) and overall survival (OS).

DETAILED DESCRIPTION:
Participants will be randomized 1:1 into two arms:

* Sacituzumab tirumotecan
* Pemetrexed plus Carboplatin

Participants will receive treatment until any of the criteria for discontinuation of study intervention are met.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced-stage nonsquamous non-small cell lung cancer (NSCLC).
* Participants who have adverse events (AEs) due to previous anticancer therapies must have recovered to Grade ≤1 or baseline.
* Participants who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load.
* Participants with history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable.
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Predominantly squamous cell histology NSCLC.
* History of second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 3 years.
* Grade ≥2 peripheral neuropathy.
* History of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing.
* Active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease.
* Uncontrolled, or significant cardiovascular disease or cerebrovascular disease.
* Received prior radiotherapy within 2 weeks of start of study intervention, or radiation-related toxicities, requiring corticosteroids.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Received radiation therapy to the lung that is >30 Gray within 6 months of the first dose of study intervention.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Active infection requiring systemic therapy.
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Concurrent active HBV and HCV infection.
* History of allogeneic tissue/solid organ transplant.
* Participants who have not adequately recovered from major surgery or have ongoing surgical complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2028-09-12 (Estimated); Study Completion 2030-06-14 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 51 months
  Progression-Free Survival is defined as the time from randomization to the first documented disease progression per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) based on blinded independent central review (BICR) or death due to any cause, whichever occurs first. PFS for all randomized participants will be reported.
Overall Survival (OS) | Up to approximately 51 months
  Overall survival is defined as the time from randomization to death due to any cause. Overall survival for all randomized participants will be reported.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 51 months
  The objective response rate (ORR) is defined as a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by BICR. The overall response rate for all randomized participants will be reported.
Duration of Response (DOR) | Up to approximately 51 months
  For participants who demonstrate confirmed CR or PR per RECIST 1.1 as assessed by BICR, duration of response is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score | Baseline and up to approximately 6 years
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) are scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores are standardized so that scores range from 0 to 100. A higher value indicates a better level of function. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be reported.
Change From Baseline in the Dyspnea (Item 8) Score, on the EORTC QLQ-C30 | Baseline and up to approximately 6 years
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the question "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized so that scores range from 0 to 100. A higher value indicates increased severity of symptoms. Change from baseline in dyspnea (EORTC QLQ-C30 Item 8) will be reported.
Change from Baseline in the Cough (Item 31) Score, on the EORTC Lung-Cancer specific Quality of Life Questionnaire (QLQ-LC13) | Baseline and up to approximately 6 years
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher value indicates increased severity of symptoms. Change from baseline in cough (EORTC QLQ-LC13 Item 31) will be reported.
Change from Baseline in the Chest Pain (Item 40) Score, on the EORTC QLQ-LC13 | Baseline and up to approximately 6 years
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher value indicates increased severity of symptoms. Change from baseline in chest pain (EORTC QLQ-LC13 Item 40) score will be presented.
Time to Deterioration (TTD) in Global Health Status/Quality of Life (Items 29 and 30) Combined Score, on the EORTC QLQ-C30 | Baseline and up to approximately 6 years
  EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to Items 29 and 30 ("How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. TTD in Global Health Status (GHS)/Quality of Life (QoL) is defined as the time from baseline to the first onset of a ≥10-point decrease from baseline in combined GHS/QoL score. The TTD in GHS/QoL (Items 29 and 30) combined score will be reported.
TTD in the Dyspnea (Item 8) Score, on the EORTC QLQ-C30 | Baseline and up to approximately 6 years
  EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to the question for Item 8 "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). TTD is defined as the time from baseline to the first onset of a ≥10-point decrease from baseline in score. The TTD in dyspnea score (EORTC QLQ-C30 Item 8) will be reported.
TTD in the Cough (Item 31) Score, on the EORTC QLQ-LC13 | Baseline and up to approximately 6 years
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question for Item 31 "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). TTD is defined as the time from baseline to the first onset of a ≥10-point decrease from baseline in score. The TTD in cough score (EORTC QLQ-C30 Item 31) will be reported.
TTD in the Chest Pain (Item 40) Score, on the EORTC QLQ-LC13 | Baseline and up to approximately 6 years
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question for Item 40 "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. TTD is defined as the time from baseline to the first onset of a ≥10-point decrease from baseline in score. The TTD in chest pain score (EORTC QLQ-C30 Item 40) will be reported.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 6 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience one or more AEs will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 6 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (155):
- United States (16):
  - Kaiser Permanente - Oakland ( Site 0054), Oakland, California
  - Kaiser Permanente - Roseville ( Site 0055), Roseville, California
  - Kaiser Permanente - San Francisco ( Site 0056), San Francisco, California
  - Kaiser Permanente - Santa Clara ( Site 0057), Santa Clara, California
  - Kaiser Permanente-Kaiser Permanente ( Site 0036), Vallejo, California
  - Kaiser Permanente - Walnut Creek ( Site 0058), Walnut Creek, California
  - Mid Florida Hematology and Oncology Center ( Site 0005), Orange City, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 0003), Marietta, Georgia
  - University of Michigan ( Site 0009), Ann Arbor, Michigan
  - Cox Medical Center North - Cox Medical Center/ Hematology/Medical Oncology ( Site 0051), Springfield, Missouri
  - Astera Cancer Care ( Site 0032), East Brunswick, New Jersey
  - Stony Brook University-Cancer Center ( Site 0038), Stony Brook, New York
  - Sanford Fargo Medical Center ( Site 0028), Fargo, North Dakota
  - Sanford Cancer Center ( Site 0024), Sioux Falls, South Dakota
  - University of Texas MD Anderson ( Site 0063), Houston, Texas
  - Millennium Research & Clinical Development ( Site 0035), Houston, Texas
- Argentina (6):
  - Clinica Adventista Belgrano-Oncology ( Site 0315), Caba., Buenos Aires
  - Instituto Alexander Fleming ( Site 0307), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Británico de Buenos Aires-Oncology ( Site 0304), Buenos Aires, Buenos Aires F.D.
  - Centro Privado de RMI Río Cuarto S.A. II ( Site 0310), Río Cuarto, Córdoba Province
  - Instituto de Oncología de Rosario ( Site 0301), Rosario, Santa Fe Province
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 0303), La Rioja
- Canada (4):
  - Cross Cancer Institute ( Site 0201), Edmonton, Alberta
  - Waterloo Regional Health Network (WRHN) ( Site 0207), Kitchener, Ontario
  - Princess Margaret Cancer Centre ( Site 0203), Toronto, Ontario
  - McGill University Health Centre ( Site 0204), Montreal, Quebec
- China (26):
  - Anhui Provincial Cancer Hospital ( Site 3132), Hefei, Anhui
  - Beijing Cancer hospital ( Site 3100), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-pneumology department ( Site 3107), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital-Medical Oncology ( Site 3128), Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital ( Site 3124), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 3125), Xiamen, Fujian
  - Southern Medical University Nanfang Hospital-Depatrment of Respiratory and Critical Care Medicine ( Site 3102), Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital-Respiratory Oncology ( Site 3103), Nanning, Guangxi
  - Harbin Medical University Cancer Hospital ( Site 3109), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 3105), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 3121), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 3122), Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University-Oncology ( Site 3104), Changsha, Hunan
  - Nanjing Drum Tower Hospital JiangBei International Branch Hospital ( Site 3117), Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University-Respiratory Department ( Site 3118), Suzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University ( Site 3119), Nanchang, Jiangxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University ( Site 3130), Xi'an, Shaanxi
  - Jinan Central Hospital ( Site 3113), Jinan, Shandong
  - Shandong Cancer Hospital ( Site 3112), Jinan, Shandong
  - Zhongshan Hospital of Fudan University ( Site 3133), Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital ( Site 3114), Taiyuan, Shanxi
  - West China Hospital, Sichuan University ( Site 3126), Chengdu, Sichuan
  - Sichuan Cancer hospital. ( Site 3127), Chengdu, Sichuan
  - The first Affiliated Hospital, Zhejiang University School of Medicine ( Site 3101), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine-Medical Oncology ( Site 3106), Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Respiratory department ( Site 3120), Wenzhou, Zhejiang
- Colombia (6):
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0600), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 0606), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 0601), Valledupar, Cesar Department
  - IMAT S.A.S ( Site 0602), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 0604), Pereira, Risaralda Department
  - Fundacion Valle del Lili- CIC-Oncology CIC ( Site 0605), Cali, Valle del Cauca Department
- France (4):
  - Nouvel Hôpital Civil (NHC) ( Site 1302), Strasbourg, Alsace
  - Clinique Clairval ( Site 1306), Marseille, Bouches-du-Rhone
  - Hopitaux Universitaires Paris Centre-Hopital Cochin-Unité d'Oncologie Thoracique ( Site 1304), Paris
  - Gustave Roussy ( Site 1303), Villejuif, Île-de-France Region
- India (6):
  - Artemis hospital ( Site 3307), Gurugram, Haryana
  - Tata Memorial Hospital-Medical Oncology ( Site 3304), Mumbai, Maharashtra
  - Kokilaben Dhirubhai Ambani Hospital & Medical Research Institute-Centre for cancer ( Site 3302), Mumbai, Maharashtra
  - All India Institute of Medical Sciences-Department of medical oncology ( Site 3303), New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospitals-APOLLO RESEARCH INNOVATION ( Site 3301), New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute And Research Centre ( Site 3300), New Delhi, National Capital Territory of Delhi
- Italy (5):
  - Instituto Tumori Giovanni Paolo II-SSD Oncologia Medica per la Patologia Toracica ( Site 1802), Bari, Apulia
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1800), Milan, Lombardy
  - Istituto Europeo di Oncologia IRCCS-Divisione di Oncologia Toracica ( Site 1803), Milan, Lombardy
  - Azienda Ospedaliera Universitaria Careggi-SOD ONCOLOGIA MEDICA ( Site 1804), Florence, Tuscany
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 1801), Roma
- Japan (19):
  - Fujita Health University Hospital ( Site 3409), Toyoake, Aichi-ken
  - Ehime University Hospital ( Site 3411), Tōon, Ehime
  - National Hospital Organization Kyushu Cancer Center ( Site 3401), Fukuoka, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 3413), Ōta, Gunma
  - Kanazawa University Hospital ( Site 3402), Kanazawa, Ishikawa-ken
  - St. Marianna University Hospital ( Site 3415), Kawasaki, Kanagawa
  - Kanagawa Cancer Center ( Site 3416), Yokohama, Kanagawa
  - Miyagi Cancer Center ( Site 3406), Natori-shi, Miyagi
  - Kansai Medical University Hospital ( Site 3414), Hirakata, Osaka
  - Saitama Prefectural Cancer Center ( Site 3417), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center ( Site 3405), Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 3408), Chūō, Tokyo
  - Toho University Omori Medical Center ( Site 3407), Ōta-ku, Tokyo
  - Kyushu University Hospital ( Site 3400), Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital ( Site 3419), Hiroshima
  - Niigata Cancer Center Hospital ( Site 3403), Niigata
  - Okayama University Hospital ( Site 3404), Okayama
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 3410), Osaka
  - Osaka Metropolitan University Hospital ( Site 3412), Osaka
- Malaysia (5):
  - University Malaya Medical Centre ( Site 3507), Lembah Pantai, Kuala Lumpur
  - National Cancer Institute-Radiotherapy and Oncology ( Site 3504), Putrajaya, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan ( Site 3506), Kuantan, Pahang
  - Hospital Pulau Pinang-Oncology, radiotherapy and palliat ( Site 3501), George Town, Pulau Pinang
  - Sarawak General Hospital-Radiotherapy Unit ( Site 3508), Kuching, Sarawak
- Mexico (5):
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 0700), Guadalajara, Jalisco
  - Arké SMO S.A. de C.V. ( Site 0706), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Servicio de Oncología ( Site 0705), Monterrey, Nuevo León
  - Oaxaca Site Management Organization S.C. ( Site 0701), Oaxaca City
  - Centro de Investigacion Clinica de Oaxaca ( Site 0704), Oaxaca City
- Poland (4):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 2003), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 2000), Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii ( Site 2010), Bialystok, Podlaskie Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach-II Klinika Radioterapi i Chemioterapii ( Site 2002), Gliwice, Silesian Voivodeship
- South Korea (13):
  - National Cancer Center ( Site 3803), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 3807), Seongnam, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital ( Site 3800), Suwon, Kyonggi-do
  - Ajou University Hospital ( Site 3813), Suwon, Kyonggi-do
  - Pusan National University Yangsan Hospital ( Site 3802), Pusan, Kyongsangnam-do
  - Chungbuk National University Hospital ( Site 3804), Cheongju-si, North Chungcheong
  - Pusan National University Hospital ( Site 3805), Busan, Pusan-Kwangyokshi
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 3814), Daegu, Taegu-Kwangyokshi
  - Chungnam national university hospital ( Site 3806), Junggu, Taejon-Kwangyokshi
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital ( Site 3812), Seoul
  - Asan Medical Center ( Site 3810), Seoul
  - Samsung Medical Center ( Site 3811), Seoul
  - Korea University Guro Hospital ( Site 3808), Seoul
- Spain (4):
  - Institut Català d'Oncologia - L'Hospitalet-Medical Oncology ( Site 2321), LHospitalet de Llobregat, Barcelona
  - CHUS - Hospital Clinico Universitario-Servicio de Oncologia ( Site 2322), Santiago de Compostela, La Coruna
  - Hospital Universitario Juan Ramon Jimenez-Oncología Medica ( Site 2323), Huelva
  - Hospital Universitario Virgen Macarena-Unidad de Investigación Oncológica ( Site 2324), Seville
- Karolinska Universitetssjukhuset Solna ( Site 2401), Stockholm, Stockholm County, Sweden
- Taiwan (12):
  - National Cheng Kung University Hospital ( Site 3901), Tainan, Tainan
  - Chi Mei Hospital - Liouying Branch ( Site 3909), Tainan, Tainan
  - National Taiwan University Cancer Center (NTUCC) ( Site 3907), Taipei City, Taipei
  - Changhua Christian Hospital ( Site 3904), Changhua
  - National Taiwan University Hospital - Hsinchu branch ( Site 3900), Hsinchu
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 3905), Kaohsiung City
  - Far Eastern Memorial Hospital ( Site 3912), New Taipei City
  - Taichung Veterans General Hospital-Chest ( Site 3910), Taichung
  - National Taiwan University Hospital-Oncology ( Site 3908), Taipei
  - Mackay Memorial Hospital-Chest Medicine ( Site 3902), Taipei
  - Taipei Medical University Hospital ( Site 3903), Taipei
  - Chang Gung Medical Foundation-Linkou Branch-Clinic of Chest Medicine ( Site 3911), Taoyuan District
- Thailand (7):
  - Faculty of Medicine Siriraj Hospital ( Site 4004), Bangkok, Bangkok
  - Bangkok Metropolitan Administration Medical College and Vajira Hospital ( Site 4006), Dusit, Bangkok
  - Faculty of Medicine - Khon Kaen University ( Site 4002), Muang, Changwat Khon Kaen
  - Lampang Cancer Hospital ( Site 4000), Lampang, Changwat Lampang
  - Ramathibodi Hospital ( Site 4001), Ratchathewi, Changwat Ratchaburi
  - Songklanagarind hospital ( Site 4003), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 4005), Muang, Chiang Mai
- Turkey (Türkiye) (5):
  - Adana Medical Park Seyhan Hastanesi-Medikal Onkoloji ( Site 2504), Adana
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 2501), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 2505), Ankara
  - Ankara Bilkent Şehir Hastanesi ( Site 2500), Ankara
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 2503), Izmir
- Vietnam (7):
  - Hanoi Oncology Hospital ( Site 4198), Hanoi, Hanoi
  - K Hospital - National Cancer Hospital ( Site 4193), Hanoi, Hanoi
  - National Lung Hospital-Oncology Department ( Site 4194), Hanoi, Hanoi
  - Oncology Hospital ( Site 4191), Ho Chi Minh City, Ho Chi Minh
  - Thong Nhat Hospital ( Site 4192), Tan Binh District, Ho Chi Minh
  - Cho Ray Hospital ( Site 4190), Ho Chi Minh City
  - Tam Anh TP.HCM General Hospital ( Site 4196), Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information. — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26307&tenant=MT_MSD_9011